CLINICAL TRIAL: NCT01974453
Title: RAdiation Dose In percutANeuos Coronary Procedures Through Transradial Approach (RADIANT Observational Study)
Acronym: RADIANT
Status: Completed | Type: Observational
Sponsor: Ospedale Sandro Pertini, Roma (Other)
Responsible Party: Principal Investigator, Alessandro Sciahbasi, MD, MD, Ospedale Sandro Pertini, Roma
Other Study IDs: Pertini3
Record Dates: First submitted 2013-10-26; First posted 2013-11-01 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Radiation Exposure
Keywords: Radiation dose, transradial approach, percutaneous coronary interventions, coronary angiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day

GROUPS / COHORTS (3):
- Right transradial: Procedures performed through right transradial approach
  Interventions: Radiation: Radiation dose
- Left transradial: Procedures performed through left transradial approach
  Interventions: Radiation: Radiation dose
- Femoral: Procedures performed through transfemoral approach
  Interventions: Radiation: Radiation dose

INTERVENTIONS:
Radiation: Radiation dose — Radiation dose adsorbed by operators

SUMMARY:
Radiation issue during percutaneous coronary interventions is an important issue for operators due to the long term stochastic risk of cancer induction, but is often under-evaluated. Many factors may be associated with the radiation dose adsorbed by operators. In particular the most important are the position taken by the operator, the use of dedicated X-ray shield and the duration of the procedure. However other factors (as operator height or the angulation of the radiation tube) might have some important effects but are often under-evaluated .

Aim of our observational study is to evaluate the most important determinants of the radiation dose adsorbed by operators during different coronary procedures (diagnostic coronary angiography or percutaneous coronary interventions) and through different vascular accesses (right or left transradial approach or transfemoral approach).

All patients who underwent to percutaneous coronary diagnostic or interventional procedures will be enrolled in this observational study.

Each operator will be equipped with dedicated dosimeters placed at left wrist, at thorax level outside the lead apron and at head level to evaluate the radiation dose at crystalline. Effective doses delivered to patients will be expressed as dose area product (DAP) and measured in Gycm2.

ELIGIBILITY:
Inclusion Criteria:

All patients who underwent to percutaneous coronary diagnostic or interventional procedures

Exclusion Criteria:

hemodynamic instability, age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medical operators that performe diagnostic and interventional coronary procedures
Sampling Method: Probability Sample
Enrollment: 2028 (Actual)
Dates: Start 2012-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Radiation Dose adsorbed by operators | Periprocedural
  Radiation Dose adsorbed by operators

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Sandro Pertini - ASL RMB, Rome, RM, Italy